CLINICAL TRIAL: NCT06896448
Title: Innovative OSA Screening in Head and Neck Cancer Patients With the Apneal App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Mitral (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-0233
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS); Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with head and neck cancers (Experimental)
  Interventions: Diagnostic Test: Specialized sleep consultation and overnight recording using the APNEAL application

INTERVENTIONS:
Diagnostic Test: Specialized sleep consultation and overnight recording using the APNEAL application — A sleep consultation with a clinical examination. Completion of several questionnaires: Snoring and sleep quality questionnaire (AFSORL), EORTC Qulity of Life questionnary -C30, and H&N35.
  Providing the Apneal application pre-installed on a loaned smartphone for the patient to use at home for overnight recording.

SUMMARY:
Obstructive sleep apnea syndrome is a common but often underdiagnosed condition, with significant impacts on quality of life, such as fatigue, attention disorders, and an increased risk of heart attack or stroke. Structural changes in the head and neck region appear to contribute to the onset or worsening of this condition.

To improve patients' quality of life, early diagnosis is essential. Currently, diagnosis relies on expensive devices, often associated with long waiting times. To address these challenges, an innovative solution is proposed: a smartphone application enabling a simple and accessible diagnosis. This application is currently under validation and has not yet been commercialized.

The purpose of the study is to determine whether this smartphone application can be used in clinical practice for patients with a head and neck lesion to diagnose sleep apnea syndrome and to assess its progression during the medical care. This study is for patients who present a head and neck lesion currently under evaluation in our department at Caen University Hospital.

This research will be integrated into routine follow-up for a period of six months.

The medical device used in this study, Apneal, is a smartphone application currently undergoing validation for the rapid diagnosis of sleep apnea syndrome. Its use is simple: the smartphone is placed in airplane mode and secured to the chest overnight. Using the phone's built-in sensors, respiratory sleep data is collected and analyzed.

As part of the initial assessment, a dedicated sleep consultation is included, during which a few questionnaires are completed, followed by an overnight sleep recording using the Apneal application. This will be conducted at the beginning of the care during the assessment phase and again six months after the completion of any potential treatment.

Depending on the results, if they are inconclusive, an additional sleep recording may be required using a ventilatory polygraphy device.

This study involves only two overnight recordings with a smartphone secured to the chest, which we will set up during the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing diagnostic workup for a lesion suspected to be a head and neck cancer, followed by confirmation of the malignant nature of the lesion. The following locations will be included: the nasopharynx, nasal cavities, sinuses, oral cavity, oropharynx, hypopharynx, larynx, and parotid gland.
* The collection of the informed consent signature is required.
* The patient must be affiliated with the social security system.

Exclusion Criteria:

* Minor patients, or those under judicial protection, guardianship, or curators.
* Lack of confirmation of the malignant nature of the lesion.
* Diagnosis of metastatic cancer.
* Known history of obstructive sleep apnea syndrome (OSAS) or previously treated head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of the rate of usable collected data at 6 months after treatment, with an interim analysis after the first consultation and initial recording, meaning a given Apnea-Hypopnea Index (AHI) from at least 6 hours of overnight recording | 8 months
  Study the feasibility of screening for obstructive sleep apnea syndrome (OSAS) in clinical practice among patients with head and neck cancer using the Apneal application, which is currently under validation The patient is treated during around 2 months and the night recording will be at 3 and 6 months after the end of the treatment The number of the recording nights with at least 4 hours records will be calculated

SECONDARY OUTCOMES:
Measurement of the evolution of the AHI score during patient management, comparing the first recording with the second one performed six months after treatment completion | 8 months
  Study the incidence of obstructive sleep apnea syndrome (OSAS) in patients treated for head and neck cancer, based on the therapeutic strategy used, to identify patient profiles at higher risk of developing OSAS The IHA score will be compared
  IHA score :
  < 5 : no OSAS 5-15 : mild OSAS 15-30 : moderate OSAS > 30 : severe OSAS
  First recording at the inclusion, then 2 months of treatment and 6 months after the end of the treatment, another recording
Measurement of the evolution of quality of life criteria by comparing the initial questionnaires completed during the first consultation with those completed 6 months after treatment | 8 months
  Study the impact of obstructive sleep apnea syndrome (OSAS) on the quality of life in patients treated for head and neck cancer with the EORTC QLQ H&N35

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, France, France

IPD SHARING:
Plan to Share IPD: No